CLINICAL TRIAL: NCT01421095
Title: Ovarian Reserve Testing in Female Young Adult Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Hui-Chun Irene Su, Assistant Professor of Reproductive Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ORT study
Record Dates: First submitted 2011-06-15; First posted 2011-08-22 (Estimated); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Infertility
Keywords: Fertility; adolescent; young adult; cancer survivors
MeSH Terms: conditions — Neoplasms; Infertility | interventions — follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Basal Testing (Experimental)
  Interventions: Drug: recombinant FSH

INTERVENTIONS:
Drug: recombinant FSH — Each participant will recieve recombinant FSH (150 IU) intravenously
  Other Names: Gonal F

SUMMARY:
Young adult cancer survivors constitute an under served population to whom fertility potential is particularly important. For female young adult patients, cancer treatment such as alkylating chemotherapy are toxic to the finite number of eggs they have, resulting in risks of infertility and premature menopause related to ovarian failure. Reproductive issues are a major concern for young cancer survivors, but one that is understudied. Young cancer survivors have few tools to measure post-treatment ovarian reserve, or the quantity and quality of remaining eggs4. Accurate determination of ovarian reserve and fertility potential would not only be an important research tool, but also directly impact clinical management. The purpose of this study is to test if basal and provocative ovarian reserve testing can predict return of menses in female young adult cancer survivors, to compare basal and provocative ovarian reserve testing results between female young adult cancer survivors and healthy controls, and to compare basal and provocative ovarian reserve testing results between female young adult cancer survivors on and off of combined estrogen and progesterone hormone products.

Participants will be asked to keep track of their periods over three months. If a participant is taking birth control pills, patches, or vaginal ring, they will asked to come off the birth control for 3 months. Participants will also be asked to undergo ovarian reserve testing by blood draws and pelvic ultrasounds at the start and end of the 3 months.

DETAILED DESCRIPTION:
Same as brief summary

ELIGIBILITY:
Inclusion Criteria:

* Postmenarchal
* Cancer diagnosis
* Prior exposure to gonadotoxic therapy, inclusive of chemothearpy, pelvic or total body irradiation, unilateral oophorectomy
* A minimum of 1 year since completion of gonoadotoxic therapy
* Intact uterus
* At least one ovary

Exclusion Criteria:

* Estrogen receptor positive cancers

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2011-01-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Return of menses | 3 months
  Self reported via bleeding calenders

SECONDARY OUTCOMES:
Blood levels of FSH | 3 months
Blood levels of estradiol | 3 months
Blood levels of AMH | 3 months
Blood levels of inhibin B | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: H. Irene Su, MD MSCE, Principal Investigator — UC San Diego
Locations (1):
- UCSD Moores Cancer Center, San Diego, California, United States